CLINICAL TRIAL: NCT05255809
Title: Effects of Alexander Technique In Addition To Routine Physical Therapy On Balance, Posture And Functional Mobility In Chronic Hemorrhagic Stroke: A Randomised Controlled Trial
Brief Title: Alexander Technique, Routine Physical Therapy, Balance, Posture, Functional Mobility , Chronic, Hemorrhagic, Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Kaneez Fatima, Effects of Alexander Technique In Addition To Routine Physical Therapy On Balance, Posture And Functional Mobility In Chronic Hemorrhagic Stroke: A Randomized Controlled Trial, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/1087/2021
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Chronic Hemorrhagic Stroke
Keywords: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alexander Technique + Routine Physical Therapy (Experimental): Routine Physical Therapy+Alexander Technique Verbal Instructions in Trunk stabilising exercises. The time duration will be 15 minutes. Verbal instructions in Stance Phase Time duration 15 minutes.Ankle Strategy. 40 minutes with rest of 5 minutes after 10 minutes. Lessons would be two days a week for 16 weeks.
  Interventions: Other: Alexander Technique + Routine Physical Therapy; Other: Routine Physical Therapy
- Control Group (Placebo Comparator): Routine Physical Therapy duration: two days a week for 16 weeks. Trunk stabilising exercises time duration will be 15 minutes. Stance Phase time duration will be 15 minutes.Ankle Strategy. 40 minutes with rest of 5 minutes after 10 minutes.
  Interventions: Other: Routine Physical Therapy

INTERVENTIONS:
Other: Alexander Technique + Routine Physical Therapy — Verbal Instructions in Trunk stabilizing exercises. The time duration will be 15 minutes. Verbal instructions in Stance Phase Time duration 15 minutes.Ankle Strategy. 40 minutes with rest of 5 minutes after 10 minutes. Lessons would be two days a week for 16 weeks.
  Arms: Alexander Technique + Routine Physical Therapy
Other: Routine Physical Therapy — Trunk stabilising exercises time duration will be 15 minutes. Stance Phase time duration will be 15 minutes. Ankle Strategy. 40 minutes with rest of 5 minutes after 10 minutes. Two days a week for 16 weeks.

SUMMARY:
MATERIALS AND METHODS Design: The randomized controlled trial. Setting: Nusrat Abdul Rauf Centre for Enablement, Faisalabad. Sample size:40 in each group. Experimental group: Recieve Alexander Technique with Routine Physical Therapy. Control Group: Recieve Routine Physical Therapy.

DETAILED DESCRIPTION:
Control Group: Routine Physical Therapy duration: two days a week for 16 weeks.

Trunk stabilising exercises time duration will be 15 minutes,

Straight static standing.Time duration 15 minutes. Shoulders extend. Threestepsfeet placement.10cm away. Open eye target at 2m away. Arms by side.

Ankle Strategy. 40 minutes with rest of 5 minutes after 10 minutes. Raise heel with straight foot & straight head. 20 minutes. Foot raise with straight foot & straight head. 20 minutes. Rest.5 minutes.

Experimental Group: Alexander Technique + Routine Physical Therapy duration for two days a week for 16 weeks. Lessons will be 32.

Verbal Instructions in Trunk stabilising exercises. Lift the lumber, Head in Centre, fix hands and feet. The time duration will be 15 minutes,

Verbal instructions in Stance Phase:

Relax-Lighten up-Relax-Pull-up. "Shoulder back", "head up", "tummy in" and "stand up straight".

Hip and feet width apart.

Straight static standing.Time duration 15 minutes. Shoulders extend. Threestepsfeet placement.10cm away. Open eye target at 2m away. Arms by side.

Ankle Strategy. 40 minutes with rest of 5 minutes after 10 minutes. Raise heel with straight foot & straight head. 20 minutes. Foot raise with straight foot & straight head. 20 minutes. Rest.5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Hemorrhagic Hemiplegic Stroke.
* Age40-60Yrs.
* Both genders.
* Intact cognition by MMSE.
* Muscle tone assessment by Ashworth scale.
* Right or left side.
* 6th month onset. Exclusion Criteria: -
* Dizziness.
* Vertigo.
* Cerebellum damage.
* Hearing impairment.
* Vision impairment

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-09-29 (Estimated); Study Completion 2022-10-10 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | 16 week
  The balance will be assessed by the Berg balance scale includes fourteen items .(0-20) specifies high fall risk. (21-50) specifies medium fall risk. (41-56) specifies low fall risk.
Postural Assessment Scale for Stroke | 16 week
  The postural assessment scale for stroke comprised 12 items with a score range of 36. Static and Dynamic PASS rate from 0-3 0 indicates the lowest level of function and 3 indicates the highest level of function.
Time Up and Go Test | 16 week
  Time up and Go test for measuring Distance of Walking within 10-15 seconds .

CONTACTS AND LOCATIONS:
Overall Officials: Kaneez Fatima, MS PTN*, Principal Investigator — University of Lahore
Locations (1):
- NACE, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen RG, Gurfinkel VS, Kwak E, Warden AC, Horak FB. Lighten Up: Specific Postural Instructions Affect Axial Rigidity and Step Initiation in Patients With Parkinson's Disease. Neurorehabil Neural Repair. 2015 Oct;29(9):878-88. doi: 10.1177/1545968315570323. Epub 2015 Feb 9. PMID 25665828
- [Background] Kim S. Exploring the field application of combined cognitive-motor program with mild cognitive impairment elderly patients. J Exerc Rehabil. 2018 Oct 31;14(5):817-820. doi: 10.12965/jer.1836418.209. eCollection 2018 Oct. PMID 30443528
- [Background] Kal E, van den Brink H, Houdijk H, van der Kamp J, Goossens PH, van Bennekom C, Scherder E. How physical therapists instruct patients with stroke: an observational study on attentional focus during gait rehabilitation after stroke. Disabil Rehabil. 2018 May;40(10):1154-1165. doi: 10.1080/09638288.2017.1290697. Epub 2017 Feb 24. PMID 28637152
- [Background] Becker JJ, Copeland SL, Botterbusch EL, Cohen RG. Preliminary evidence for feasibility, efficacy, and mechanisms of Alexander technique group classes for chronic neck pain. Complement Ther Med. 2018 Aug;39:80-86. doi: 10.1016/j.ctim.2018.05.012. Epub 2018 May 23. PMID 30012397